CLINICAL TRIAL: NCT03460067
Title: Selective Use of Observation After Lumpectomy and Sentinel Lymph Node Biopsy in Her-2 Positive Patients With Pathologic Complete Response to Neoadjuvant Chemotherapy
Brief Title: Omission of Radiation in Patients With Her-2 Positive Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2017-MM-BRST-Her2noRT
Record Dates: First submitted 2018-02-24; First posted 2018-03-09 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: HER2-positive Breast Cancer
Keywords: omission of radiation; trastuzumab; pertuzumab; biospecimen collection; lumpectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Arm A (Experimental): Patient is required to have lumpectomy with sentinel lymph node biopsy shows pCR and will complete 1 year of trastuzumab +/- pertuzumab treatment. No radiation, or an omission of radiation, will be given on this arm, including external beam, brachytherapy or intraoperative radiation. Patients will be required to follow up with a medical, surgical, or radiation oncologist every 3 months for 5 years. At these follow up visits, a physical exam will be performed to assess for any disease recurrence. Screening mammogram or MRI is recommended every 6 months for patients on this arm.
  Interventions: Radiation: Omission of Radiation
- Arm B (No Intervention): Patient is required to have her-2 positive breast cancer, clinically node negative from exam. Patient will complete neoadjuvant chemotherapy per Medical Oncologist. This arm will undergo lumpectomy with sentinel lymph node biopsy shows pCR. The patient will proceed with radiation as standard of care. This arm includes a review of outcomes in the patient's medical chart as well as a collection of biospecimens such as blood and urine, for correlative studies.
- Arm C (No Intervention): Patient is required to have her-2 positive breast cancer, clinically node negative from exam. patient will complete neoadjuvant chemotherapy per Medical Oncologist. This arm will not undergo lumpectomy with sentinel lymph node biopsy shows pCR. The patient will proceed with radiation as standard of care. This arm includes a review of outcomes in the patient's medical chart as well as a collection of biospecimens, such as blood and urine, for correlative studies.

INTERVENTIONS:
Radiation: Omission of Radiation — No Radiation will be given. 1 year of trastuzumab +/- pertuzumab treatment will be given with 5 years of follow up occurring every 3 months to check for recurrence
  Arms: Arm A

SUMMARY:
The primary objective of this study is to describe the rate of local control in patients with her-2 positive early stage breast cancer with a complete response to chemotherapy and lumpectomy alone.

DETAILED DESCRIPTION:
Participants, ages 40 and older diagnosed with stage I or stage II her-2 positive, node negative breast cancer patients will be recommended to continue trastuzumab +/- pertuzumab therapy after surgery to complete a full year of therapy as standard of care under the clinical management of the patient's medical oncologist.

Once neoadjuvant chemotherapy has been completed, the patient will be separated in to one of three arms based on a set of criteria for each. If the patient wishes to take part in the study, but does not have a lumpectomy with sentinel lymph node biopsy showing pCR, the patient will be placed in to Arm C and will proceed with radiation as standard of care. If the patient wishes to take part in the study, and has a lumpectomy with sentinel lymph node biopsy showing pCR, but does not agree to omission of radiation, the patient will be placed in to Arm B and will proceed with radiation as standard of care. If the patient wishes to take part in the study, and has a lumpectomy with sentinel lymph node biopsy showing pCR and agrees to omission of radiation, the patient will be placed in to Arm A with follow up assessments occuring at 1 month post-op, and every 3 months up to 5 years post-op.

Data will be collected on local, regional and distant recurrence at each follow-up.The self-administered FACT-B+4 quality of life questionnaire will be given to patients at baseline, at first postoperative visit, and at the one year post-operative visit.

Patients enrolling prior to chemotherapy will be asked to fill out the Breast-Q™ at the time of their first surgical consultation. Patients enrolled post-surgery will be asked to fill out the Breast-Q™ at their first post-operative visit. All patients will be asked to fill out the Breast-Q™ at their yearly postoperative visits. The Breast-Q™ is a validated patient assessment of breast cosmesis. This tool has both pre operative and post-operative components. Pre-operative Breast-Q™ questionnaire data is not required of participants in this study who enroll postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent.
* Karnofsky Performance Status 50% to 100% (Appendix A).
* Women 40 years of age or older with a diagnosis of invasive ductal carcinoma
* Her-2 3+ or FISH ratio of 2.2 or higher, background gene expression with normal copy number
* Only postmenopausal women will be eligible. Subjects will be classified as being postmenopausal if they have had:

  * No spontaneous menses > 1 year, or
  * Bilateral surgical oophorectomy, or
  * No menses for < 1 year with FSH and estradiol levels in according to institutional standards
* cT1-2N0 on clinical staging (verified to have no suspicious axillary or internal mammary nodes on MRI or ultrasound)
* Undergo neoadjuvant chemotherapy with a trastuzumab based regimen prior to surgery and plan for completion of one year of trastuzumab
* Patients are required to undergo lumpectomy with sentinel lymph node biopsy
* Pathologic review shows no evidence of residual disease in the tumor bed (to also include no evidence of residual DCIS)
* Tumor bed should be no larger than 5 cm in size on pathologic review
* Fibrotic area of prior tumor located at least 3 mm away from surgical margins
* No evidence of treatment related change in the lymph nodes on pathologic review

Exclusion Criteria

* Diagnosis of inflammatory breast cancer
* Previously diagnosed malignancy excluding basal or squamous cell carcinoma of the skin (unless disease-free for 5 years or more)
* Diagnosis of metastatic disease

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2027-07-16 (Estimated); Study Completion 2027-07-16 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral Breast Cancer Recurrence | up to 5 year post-op
  Defined as biopsy positive her-2 positive tumor in the same breast

SECONDARY OUTCOMES:
Regional Nodal Recurrence | 1 month post-op, every three months post-op for 5 years
  Will include recurrence in the ipsilateral draining axilla, supraclavicular fossa, or internal mammary nodes.
Distance Metastasis | 1 month post-op, every three months post-op for 5 years
  Defined as biopsy proven disease outside of the affected breast and draining lymphatics, or definitive radiographical evidence of distant disease, to include a positive bone scan or enhancing lesions on MRI brain.
Overall Survival | 1 month post-op, every three months post-op for 5 years
  Defined as death from any cause
Quality of Life using FACT-B+4 | 1 month post-op, every three months post-op for 5 years
  Measured using scores from patient reported outcomes from FACT-B+4 questionnaire
Cosmetic (Breast) Outcomes | 1 month post-op, every three months post-op for 5 years
  Measured using scores from patient reported outcomes using the Breast Q questionnaire
Lymphedema Rate | 1 month post-op, every three months post-op for 5 years
  Assessed by a diagnosis of Lymphedema in the medical record by trained lymphedema nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Shane Stecklein, MD, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center/ Cancer Center, Kansas City, Kansas, United States